CLINICAL TRIAL: NCT00386451
Title: Prospective Study Which Compares the Use of a Closing System Without a Needle and With Positive Pressure to a Heparin Lock With Positive Pressure for Patients With a Catheter for Chemotherapy
Brief Title: Comparing a Closing System Without a Needle With Positive Pressure to a Heparin Lock With Positive Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Caren Randon, University Hospital Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/331
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Neoplasms
Keywords: Intravenous chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Catheter locking systems

SUMMARY:
A prospective randomized study to compare 2 groups:

* heparine lock with positive pressure
* lock without a needle with positive pressure

ELIGIBILITY:
Inclusion Criteria:

* Oncological patients who require intravenous chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Caren Randon, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be